CLINICAL TRIAL: NCT05866302
Title: Parametric Response Mapping (PRM) for the Detection of Chronic Lung Injury in Hematopoietic Cell Transplant Recipients. A Multi-center, Observational Trial.
Brief Title: Parametric Response Mapping (PRM) for the Detection of Chronic Lung Injury in Hematopoietic Cell Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UMCC 2022.052; HUM00225273 (Other: University of Michigan); R01HL162661 (NIH)
Record Dates: First submitted 2023-04-13; First posted 2023-05-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lung Disease; Hematopoietic Cell Transplantation; Graft Versus Host Disease
Keywords: Parametric response mapping
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be processed and shipped to an outside lab.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Newly diagnosed chronic GVHD: All subjects will undergo a non-contrast, high resolution CT scan with inspiratory and expiratory imaging, pulmonary function testing (PFT) and serologic biomarker studies upon entry. A total of 300 subjects (200 adults, 100 pediatric) will be enrolled. Patients in cohort 1 who develop CLD prior to the 12-month period will transition to cohort 2 at that time. PFT is recommended every 3 months over a 12 month period. Plasma samples will be collected at entry and at 12 months.
- Cohort 2: Newly diagnosed chronic lung disease (CLD): All subjects will undergo a non-contrast, high resolution CT scan with inspiratory and expiratory imaging, pulmonary function testing (PFT) and serologic biomarker studies upon entry. A total of 75 subjects (50 adults, 25 pediatric) will be enrolled. PFT is recommended every 3 months over a 12 month period. Plasma samples will be collected at entry and at 12 months.

SUMMARY:
The study will have two separate patient cohorts: Cohort 1 will include patients with newly diagnosed chronic graft versus host disease (GVHD), whereas cohort 2 will include patients with newly diagnosed chronic lung disease (CLD). For cohort 1, the primary objective will be to characterize PRM metrics at the onset of chronic GVHD and determine if a PRM signature is present that will predict 1-year CLD free survival. For cohort 2, the primary objective will focus on characterizing PRM at the onset of CLD and determine if PRM can predict the trajectory in lung function decline in affected patients.

ELIGIBILITY:
Inclusion Criteria:

* For both Cohorts 1 and 2:
* Age ≥ 36 months. There is no upper age limit.
* Receipt of an allogeneic HCT. There are no exclusions to study entry based upon primary diagnosis, hematopoietic cell source, conditioning regimen, donor type, degree of donor-recipient HLA match, or current organ function.
* All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Cohort 1 (Chronic Graft Versus Host Disease): Diagnosis of chronic GVHD in at least 1 organ system within the prior 3 months. NIH Consensus Criteria for chronic GVHD are required to establish the diagnosis. (https://pubmed.ncbi.nlm.nih.gov/25529383/)
* Cohort 2 (Chronic Lung Disease, CLD) Diagnosis of CLD within the prior 100 days, including either Bronchiolitis Obliterans Syndrome (BOS) or Restrictive lung disease (RLD), with each defined as follows: Bronchiolitis Obliterans Syndrome (BOS): (NIH Consensus Criteria)31 a.FEV1 < 75% predicted, with a decline in absolute FEV1 > 10% compared to pretransplant baseline or within the prior 2 years, b.FEV1/VC or FEV1/FVC < 0.7 , c. Absence of an alternative diagnosis, including COPD exacerbation, asthma, and active respiratory tract infection, as determined by appropriate clinical investigations that may include chest imaging, microbiologic cultures, and/or bronchoscopy, d. One of two supportive features of BOS: i. Evidence of air trapping by PFTs: RV>120%, or elevated RV/TLC (>20% of predicted), ii. High resolution chest CT with inspiratory and expiratory cuts that show findings that are consistent with small airways disease including (but not exclusive of) air trapping, bronchial wall thickening, or bronchiectasis. Restrictive Lung Disease (RLD): a. ≥ 20% decline in FEV1 from baseline, coupled with ≥ 10% decline in total lung capacity (TLC) from baseline. If measurements of TLC are not available, then a ≥ 20% decline in FVC from baseline may be substituted for RLD.32, b.Radiographic opacities or infiltrates on chest radiograph or CT. Such changes may include, but are not limited to the presence of ground glass opacities, reticular changes, septal thickening, fibrotic changes or areas of consolidation.
* Patients unable to perform PFT. For cohort 1, patient's too young (or physically unable) to perform PFT's remain eligible provided they meet all other eligibility criteria. For cohort 2, children too young (or physically unable) to perform PFT's are eligible provided they exhibit both clinical and radiographic features (on CT) consistent with CLD. Clinical features would include dyspnea, cough, and/or SpO2 < 93% on room air. Radiographic features may include, but are not limited to the presence of air trapping, bronchial wall thickening, or bronchiectasis.

Exclusion Criteria:

* Relapse of a patient's primary malignancy post-HCT, or the development of any secondary "hematologic" malignancy post-HCT.
* The presence of an active, uncontrolled infection.
* Patients who would require intubation solely for the purposes of obtaining a CT scan for PRM imaging. (In contrast, if a clinical CT is being performed as routine medical care to evaluate a patient's lung function, the patient is eligible and PRM imaging may be performed from that CT.)

Min Age: 36 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult HCT populations
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
1-year CLD free survival (Cohort 1) | up to 12 months from enrollment
  The time to develop CLD or death over 12 months of follow-up in both pediatric and adult subjects will be determined. we will classify subjects into comparison groups of (1) high PRMfSAD (>30%), (2) high PRMPD (>40%) or (3) neither high PRMfSAD nor high PRMPD (PRMNorm group). The two primary analyses are to compare 1-year CLD-free survival between the high PRMfSAD and PRMNorm groups and separately between the high PRMPD and PRMNorm groups, using two-sided, two-sample logrank tests with an overall 5% type I error, adjusted for 2 comparisons using the Bonferroni method
FEV1 decline (Cohort 2) | up to 12 months from enrollment
  Trajectory of FEV1 decline over a 12-month period in patients with newly diagnosed CLD. To evaluate PRM as a predictor of "lung function decline" in patients with an established diagnosis of CLD.

SECONDARY OUTCOMES:
PRM profiles in children at the onset of chronic GVHD (Cohort 1) | up to 12 months from enrollment
  Pediatric subjects will be enrolled into one of 2 strata (PFT+ vs PFTnull), PRM imaging with whole lung volumetric CT scans will be performed at baseline, using low dose CT techniques in children. Strata 1 (PFT+), the occurrence of CLD will be defined using NIH Consensus Criteria for BOS, or ISHLT criteria for RLD. Stratum 2 (PFTnull), radiographic findings of obstructive or restrictive lung disease on CT, plus clinical symptoms (dyspnea, or hypoxia) will be required to establish a diagnosis of CLD, in lieu of PFTs. PRM profile will be reported as percent functional small airway disease (PRMfSAD), emphysema (PRMEmph), parenchymal lung disease (PRMPD), and normal lung parenchyma (PRMNorm), in relation to the total lung volume.
Correlate PRM profiles at the onset of chronic GVHD with overall survival post-HCT (Cohort 1) | up to 12 months from enrollment
  Subjects will be enrolled into one of 2 strata (PFT+ vs PFTnull), PRM imaging with whole lung volumetric CT scans will be performed at baseline.. For patients in strata 1 (PFT+), the occurrence of CLD will be defined using NIH Consensus Criteria for BOS, or ISHLT criteria for RLD. For patients in stratum 2 (PFTnull), radiographic findings of obstructive or restrictive lung disease (i.e. air trapping, bronchiectactic changes, interstitial fibrosis) on CT, plus clinical symptoms (dyspnea, or hypoxia) will be required to establish a diagnosis of CLD, in lieu of PFTs. Histograms of PRMfSAD, PRMPD, PRMEmph, and PRMNorm values will be displayed by pediatric stratum and overall, with means ± standard errors superimposed on the plots. PRM profile will be reported as percent functional small airway disease (PRMfSAD), emphysema (PRMEmph), parenchymal lung disease (PRMPD), and normal lung parenchyma (PRMNorm), in relation to the total lung volume.
To characterize a PRM profile for CLD in children post-HCT (Cohort 2) | up to 12 months from enrollment
  We will have approximately 90% power to detect correlations > 0.47 using 2-sided 1-sample correlation tests. This is a conservative estimate involving only the adult participants, with power increasing once pediatric participants are included in the analysis. In a secondary analysis we will use linear mixed effects models to study FEV1 predicted trajectories after CLD onset, as a function of PRM values. We will explore interactions between PRM values and time post-CLD when modeling FEV1 predicted values over time. PRM profile will be reported as percent functional small airway disease (PRMfSAD), emphysema (PRMEmph), parenchymal lung disease (PRMPD), and normal lung parenchyma (PRMNorm), in relation to the total lung volume.
To determine a PRM profile for restrictive lung disease (RLD) in adults with chronic GVHD post-HCT (Cohort 2) | up to 12 months from enrollment
  We will have approximately 90% power to detect correlations > 0.47 using 2-sided 1-sample correlation tests. This is a conservative estimate involving only the adult participants, with power increasing once pediatric participants are included in the analysis. In a secondary analysis we will use linear mixed effects models to study FEV1 predicted trajectories after CLD onset, as a function of PRM values. We will explore interactions between PRM values and time post-CLD when modeling FEV1 predicted values over time. PRM profile will be reported as percent functional small airway disease (PRMfSAD), emphysema (PRMEmph), parenchymal lung disease (PRMPD), and normal lung parenchyma (PRMNorm), in relation to the total lung volume.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - Stanford Hospital, Stanford, California
  - Emory University, Atlanta, Georgia
  - Dana Farber, Boston, Massachusetts
  - The University of Michigan Cancer Center, Ann Arbor, Michigan
  - MD Anderson, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No